CLINICAL TRIAL: NCT07043543
Title: Randomized Open Phase II Multienter Study Evaluating the Clinical Utility of Online Adaptive Radiotherapy in Bladder Cancer
Brief Title: Evaluation of the Clinical Utility of Online Adaptive Radiotherapy in Bladder Cancer (BLADAPT-GETUG V11)
Acronym: BLADAPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2024-02 BLA
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: Adaptive radiotherapy; standard radiotherapy; Tri-Modal therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental arm (Experimental): Adaptive radiotherapy +/- chemotherapy
  Interventions: Radiation: Adaptive radiotherapy
- standard arm (Active Comparator): Standard radiotherapy +/- chemotherapy
  Interventions: Radiation: standard radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy — Patient will be treated by concomitant:
  * adaptive radiotherapy 5 days a week for 4 weeks with hypofractionated irradiation 55 Gy / 20 fractions +/- pelvic inclusion 44 Gy/20 fractions (SIB).
  * chemotherapy if not contraindicated :
    * Cisplatin : 20 mg/m2/day on day 1 to day 4 and day 22 to day 25 (or 80 mg/m2 during week 1 and 4 of radiotherapy) Or
    * Gemcitabine: 80 to 100 mg/m2/week Or
    * Mitomycin C: 12 mg/m2 on day 1 only + 5FU infusion 500 mg/m2/day during 5 days on week 1 and 4 of radiotherapy (alternatively : capecitabine taken twice daily at a dose of 825 per square meter per day on the days of radiotherapy)
  Arms: experimental arm
Radiation: standard radiotherapy — Patient will be treated by concomitant:
  * standard 5 days a week for 4 weeks with hypofractionated irradiation 55 Gy / 20 fractions +/- pelvic inclusion 44 Gy/20 fractions (SIB).
  * chemotherapy if not contraindicated :
    * Cisplatin : 20 mg/m2/day on day 1 to day 4 and day 22 to day 25 (or 80 mg/m2 during week 1 and 4 of radiotherapy) Or
    * Gemcitabine: 80 to 100 mg/m2/week Or
    * Mitomycin C: 12 mg/m2 on day 1 only + 5FU infusion 500 mg/m2/day during 5 days on week 1 and 4 of radiotherapy (alternatively : capecitabine taken twice daily at a dose of 825 per square meter per day on the days of radiotherapy)
  Arms: standard arm

SUMMARY:
Trimodal therapy (TMT) consisting of transurethral resection of bladder tumors followed by radiotherapy and chemotherapy is a therapeutic alternative in patients with Muscle-Infiltrating Bladder Cancer who are inoperable or refuse surgery. One of the main challenges of TMT is the planning and delivery of radiation therapy. Indeed, the bladder is a mobile hollow organ subject to repletion, with variations in size and shape during and between radiotherapy sessions. Standard radiotherapy techniques require large planning target volume margins around the bladder, which can be responsible for irradiation of a large volume of large and small bowel with grade 2 and 3 toxicities.

Adaptive radiotherapy allows for the generation of a treatment fraction personalized to a patient's anatomical modification with margin reduction and improves the dosimetric quality of the delivered plans.

The hypothesis is that this improvement results in radiation-induced toxicity improvement.

DETAILED DESCRIPTION:
In 2023, the incidence of muscle-infiltrating bladder cancer (MIBC) in France was 14062 cases, 81% of which were in men.

The standard treatment for MIBC is cystectomy preceded by neoadjuvant chemotherapy. Trimodal therapy (TMT), consisting of transurethral resection of bladder tumors (TURBT) followed by radiotherapy (RT) and chemotherapy (CT), has emerged as a valuable therapeutic de-escalation alternative in patients who are inoperable or refuse surgery with its physical and psychological sequelae. TMT provides survival outcomes identical to cystectomy in selected patients and allows for bladder preservation in successful cases. TMT is an effective potential alternative to radical cystectomy for recurrent high-grade T1 urothelial cancer of the bladder who failed intravesical therapy.

One of the main challenges of TMT is the planning and delivery of radiation therapy. Indeed, the bladder is a mobile hollow organ subject to repletion, with variations in size and shape during radiotherapy sessions (intra-fractional movement) and between sessions (inter-fractional movement). To take into account these movements, standard radiotherapy techniques require large planning target volume (PTV) margins around the bladder, which can be responsible for irradiation of a large volume of large and small bowel with grade 2 and 3 toxicities up to 42% and 17% respectively.

Adaptive radiotherapy (ART) allows for the generation of a treatment fraction personalized to a patient's anatomical modification. While it was until recently only performed "offline", i.e. between two radiotherapy sessions, it is now possible to perform a daily customization of the radiotherapy session ("online") for a given patient to ensure optimal coverage of the target with minimized margins. ART allows PTV margins reduction for MIBC and improves therefore the dosimetric quality of the delivered plans.

The hypothesis is that the dosimetric improvement induced by ART results in radiation-induced toxicity improvement.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven muscle-infiltrating bladder cancer (de novo MIBC or after a history of non-muscle-invasive bladder cancer) or patients with initial high-grade T1 tumor showing Ta or T1 recurrence, or those with high-grade T1 after a course of intravesical biological therapy or chemotherapy;
* Age ≥ 18 years;
* Urothelial carcinoma (transitional cell carcinoma of the bladder, micropapillary, microcystic with trophoblastic differenciation) and squamous cell histological types are allowed;
* Stage T1-T4aN0M0
* TransUrethral Resection of Bladder Tumor (TURBT) and Position Emission Tomography- scanner and X-ray Computed Tomography (PET-CT) or Computed Tomography scan of thorax/abdomen/pelvis (without carcinological anomaly) within 8 weeks prior to the start of radiation therapy (if TURBT was performed more than 6 weeks before the inclusion visit, a new TURBT or, at least, a cystoscopy showing no progression, no residual tumour or regrowth must be done);
* Suitable for radiotherapy;
* Eastern Cooperative Oncology Group/World Human Organisation (ECOG/WHO) performance status from 0 to 2
* Negative pregnancy test (blood or urine), for women of childbearing age only;
* If the patient is sexually active, he/she must agree to use contraception deemed adequate and appropriate by the investigator throughout the period of study drug administration and 6 months after the end of treatment for both men and women.
* Affiliation to the French Social Security System;
* Dated, written and signed Informed consent

Exclusion Criteria:

* Prior pelvic radiation therapy;
* Patients with previous or concomitant other malignancy within the past 5 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least five years;
* Presence of endopenic stent;
* Inability to comply with the protocol;
* Grade 1 or greater baseline diarrhea;
* Uncontrolled inflammatory bowel disease (ulcerative colitis or Crohn's disease);
* Uncontrolled immune or cardiac or pulmonary disease;
* Patients whose regular follow-up is impossible for psychological, family, social or geographical reasons;
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent or to terminate the study;
* Pregnant or breast-feeding subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of the technique of adaptive radiotherapy in terms of acute Gastro-Intestinal toxicity. | from the Day 1 Radiotherapy to 3 months after the last day of Radiotherapy
  rate of patients without acute diarrhea grade ≥2

SECONDARY OUTCOMES:
Evaluation of all acute toxicities | from the Day 1 Radiotherapy to 3 months after the last day of Radiotherapy
  description of all acute toxicities according to Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0)
Evaluation of all late toxicities | from 3 months after the last day of Radiotherapy to 5 years after the last day of Radiotherapy
  description of all late toxicities according to Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0)
evaluation of quality of life specific to the cancer disease | at baseline, the last day of radiotherapy, every 3 months after the last day of radiotherapy, during first year and every 6 months then after until 3 years.
  Quality of life will be evaluated using European Organisation for Research and Treatment of Cancer - Quality Life Questionnaire (EORTC QLQ-C30)
evaluation of quality of life and of the measurements specific to the treatment of bladder cancer with muscle invasion | at baseline, the last day of radiotherapy, every 3 months after the last day of radiotherapy, during first year and every 6 months then after until 3 years.
  Quality of life will be evaluated using European Organisation for Research and Treatment of Cancer - Quality Life Questionnaire - Bladder Cancer (EORTC QLQ-BLM30)
evaluation of quality of life for patient ≥ 70 years old in order to establish a minimum standardized geriatric assessment | at baseline, the last day of radiotherapy, every 3 months after the last day of radiotherapy, during first year and every 6 months then after until 3 years.
  Quality of life will be evaluated using Geriatric COre DatasEt oncogeriatric (GCODE) for patient ≥ 70 years old
evaluation of quality of life for patient ≥ 70 years old (Specific to elderly people with cancer) | at baseline, the last day of radiotherapy, every 3 months after the last day of radiotherapy, during first year and every 6 months then after until 3 years.
  Quality of life will be evaluated using European Organisation for Research and Treatment of Cancer - Quality Life Questionnaire-Elderly (EORTC QLQ- ELD30) for patient ≥ 70 years old
assessment of disease free survival | At 3 and 5 years after the last day of Radiotherapy
  time interval from randomization to first carcinologic event as local or distant relapse or death
assessment of cystectomy free survival | At 3 and 5 years after the last day of Radiotherapy
  the time interval from randomization to cystectomy
assessment of overall survival | At 3 and 5 years after the last day of Radiotherapy
  the time interval from randomization to death from any cause
assessment of local control rate | At 3 and 5 years after the last day of Radiotherapy
  The presence of non-muscle-invasive or muscle-invasive bladder cancers evaluate by cystoscopy
assessment of the dosimetric results | during tthe radiotherapy for both arms
  Dosimetric results in terms of treatment volume coverage and Organ At Risk protection
evaluation of the impact of the adaptive process on fractions execution | during tthe radiotherapy for both arms
  Evaluation of duration of the treatment fractions (in minutes) in the two arms. Evaluation of the percentage of fractions fully delivered and the duration of physician/physicist mobilization for the adaptive process

CONTACTS AND LOCATIONS:
Overall Officials: Olivier RIOU, MD, Principal Investigator — INSTITUT REGIONAL DU CANCER DE MONTPELLIER
Locations (11):
- France (11):
  - Centre Georges François Leclerc, Dijon, Côte d'or
  - Institut du Cancer de Montpellier, Montpellier, Herault
  - Centre Eugène Marquis, Rennes, Ille et Vilaine
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire Atlantique
  - Centre Oscar Lambret, Lille, Nord
  - Centre de radiothérapie Bayard, Villeurbanne, Rhone
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - Institut Sainte Catherine, Avignon, Var
  - Centre de radiothérapie Saint-Louis, Toulon, Var
  - Hôpital Tenon, Paris, Île-de-France Region
  - Institut Curie, Saint-Cloud, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabaille M, Khalifa J, Tessier AM, Belhomme S, Crehange G, Sargos P. [A review of adaptive radiotherapy for bladder cancer]. Cancer Radiother. 2021 May;25(3):271-278. doi: 10.1016/j.canrad.2020.08.046. Epub 2021 Jan 2. French. PMID 33402293
- [Background] Fahmy O, Khairul-Asri MG, Schubert T, Renninger M, Malek R, Kubler H, Stenzl A, Gakis G. A systematic review and meta-analysis on the oncological long-term outcomes after trimodality therapy and radical cystectomy with or without neoadjuvant chemotherapy for muscle-invasive bladder cancer. Urol Oncol. 2018 Feb;36(2):43-53. doi: 10.1016/j.urolonc.2017.10.002. Epub 2017 Nov 6. PMID 29102254
- [Background] Huddart R, Hafeez S, Omar A, Alonzi R, Birtle A, Cheung KC, Choudhury A, Foroudi F, Gribble H, Henry A, Hilman S, Hindson B, Lewis R, Muthukumar D, McLaren DB, McNair H, Nikapota A, Olorunfemi A, Parikh O, Philipps L, Rimmer Y, Syndikus I, Tolentino A, Varughese M, Vassallo-Bonner C, Webster A, Griffin C, Hall E. Acute Toxicity of Hypofractionated and Conventionally Fractionated (Chemo)Radiotherapy Regimens for Bladder Cancer: An Exploratory Analysis from the RAIDER Trial. Clin Oncol (R Coll Radiol). 2023 Sep;35(9):586-597. doi: 10.1016/j.clon.2023.05.002. Epub 2023 May 9. PMID 37225552
- [Background] Hafeez S, Lewis R, Hall E, Huddart R; RAIDER Trial Management Group. Advancing Radiotherapy for Bladder Cancer: Randomised Phase II Trial of Adaptive Image-guided Standard or Dose-escalated Tumour Boost Radiotherapy (RAIDER). Clin Oncol (R Coll Radiol). 2021 Jun;33(6):e251-e256. doi: 10.1016/j.clon.2021.02.012. Epub 2021 Mar 23. No abstract available. PMID 33766502
- [Background] Kool R, Dragomir A, Kulkarni GS, Marcq G, Breau RH, Kim M, Busca I, Abdi H, Dawidek M, Uy M, Fervaha G, Cury FL, Alimohamed N, Izawa J, Jeldres C, Rendon R, Shayegan B, Siemens R, Black PC, Kassouf W. Benefit of Neoadjuvant Cisplatin-based Chemotherapy for Invasive Bladder Cancer Patients Treated with Radiation-based Therapy in a Real-world Setting: An Inverse Probability Treatment Weighted Analysis. Eur Urol Oncol. 2024 Dec;7(6):1350-1357. doi: 10.1016/j.euo.2024.01.014. Epub 2024 Feb 6. PMID 38326142
- [Background] Dahl DM, Rodgers JP, Shipley WU, Michaelson MD, Wu CL, Parker W, Jani AB, Cury FL, Hudes RS, Michalski JM, Hartford AC, Song D, Citrin DE, Karrison TG, Sandler HM, Feng FY, Efstathiou JA. Bladder-Preserving Trimodality Treatment for High-Grade T1 Bladder Cancer: Results From Phase II Protocol NRG Oncology/RTOG 0926. J Clin Oncol. 2024 Dec;42(34):4095-4102. doi: 10.1200/JCO.23.02510. Epub 2024 Sep 3. PMID 39226514
- [Background] de Haar-Holleman A, van Hoogstraten LMC, Hulshof MCCM, Tascilar M, Bruck K; BlaZIB study group; Meijer RP, Alfred Witjes J, Kiemeney LA, Aben KKH. Chemoradiation for muscle-invasive bladder cancer using 5-fluorouracil versus capecitabine: A nationwide cohort study. Radiother Oncol. 2023 Jun;183:109584. doi: 10.1016/j.radonc.2023.109584. Epub 2023 Mar 1. PMID 36863459
- [Background] Hall E, Hussain SA, Porta N, Lewis R, Crundwell M, Jenkins P, Rawlings C, Tremlett J, Sreenivasan T, Wallace J, Syndikus I, Sheehan D, Lydon A, Huddart R, James N; BC2001 Investigators. Chemoradiotherapy in Muscle-invasive Bladder Cancer: 10-yr Follow-up of the Phase 3 Randomised Controlled BC2001 Trial. Eur Urol. 2022 Sep;82(3):273-279. doi: 10.1016/j.eururo.2022.04.017. Epub 2022 May 14. PMID 35577644
- [Background] Sibolt P, Andersson LM, Calmels L, Sjostrom D, Bjelkengren U, Geertsen P, Behrens CF. Clinical implementation of artificial intelligence-driven cone-beam computed tomography-guided online adaptive radiotherapy in the pelvic region. Phys Imaging Radiat Oncol. 2020 Dec 18;17:1-7. doi: 10.1016/j.phro.2020.12.004. eCollection 2021 Jan. PMID 33898770
- [Background] Hussain MH, Glass TR, Forman J, Sakr W, Smith DC, Al-Sarraf M, Jones J, Balcerzak SP, Crawford ED, Grossman HB. Combination cisplatin, 5-fluorouracil and radiation therapy for locally advanced unresectable or medically unfit bladder cancer cases: a Southwest Oncology Group Study. J Urol. 2001 Jan;165(1):56-60; discussion 60-1. doi: 10.1097/00005392-200101000-00014. PMID 11125363
- [Background] Azria D, Riou O, Rebillard X, Thezenas S, Thuret R, Fenoglietto P, Pouessel D, Culine S. Combined chemoradiation therapy with twice-weekly gemcitabine and cisplatin for organ preservation in muscle-invasive bladder cancer: long-term results of a phase 1 trial. Int J Radiat Oncol Biol Phys. 2014 Mar 15;88(4):853-9. doi: 10.1016/j.ijrobp.2013.11.016. Epub 2013 Dec 21. PMID 24368064
- [Background] Housset M, Maulard C, Chretien Y, Dufour B, Delanian S, Huart J, Colardelle F, Brunel P, Baillet F. Combined radiation and chemotherapy for invasive transitional-cell carcinoma of the bladder: a prospective study. J Clin Oncol. 1993 Nov;11(11):2150-7. doi: 10.1200/JCO.1993.11.11.2150. PMID 8229129
- [Background] Oh KS, Soto DE, Smith DC, Montie JE, Lee CT, Sandler HM. Combined-modality therapy with gemcitabine and radiation therapy as a bladder preservation strategy: long-term results of a phase I trial. Int J Radiat Oncol Biol Phys. 2009 Jun 1;74(2):511-7. doi: 10.1016/j.ijrobp.2008.08.021. Epub 2008 Oct 30. PMID 18977098
- [Background] Kent E, Sandler H, Montie J, Lee C, Herman J, Esper P, Fardig J, Smith DC. Combined-modality therapy with gemcitabine and radiotherapy as a bladder preservation strategy: results of a phase I trial. J Clin Oncol. 2004 Jul 1;22(13):2540-5. doi: 10.1200/JCO.2004.10.070. PMID 15226322
- [Background] Caffo O, Thompson C, De Santis M, Kragelj B, Hamstra DA, Azria D, Fellin G, Pappagallo GL, Galligioni E, Choudhury A. Concurrent gemcitabine and radiotherapy for the treatment of muscle-invasive bladder cancer: A pooled individual data analysis of eight phase I-II trials. Radiother Oncol. 2016 Nov;121(2):193-198. doi: 10.1016/j.radonc.2016.09.006. Epub 2016 Oct 5. PMID 27720221
- [Background] Bruck K, Meijer RP, Boormans JL, Kiemeney LA, Witjes JA, van Hoogstraten LMC, van der Heijden MS, Donders AR, Franckena M, Uyl de Groot CA, Leliveld AM, Aben KKH, Hulshof MCCM. Disease-Free Survival of Patients With Muscle-Invasive Bladder Cancer Treated With Radical Cystectomy Versus Bladder-Preserving Therapy: A Nationwide Study. Int J Radiat Oncol Biol Phys. 2024 Jan 1;118(1):41-49. doi: 10.1016/j.ijrobp.2023.07.027. Epub 2023 Jul 28. PMID 37517601
- [Background] Pfister C, Gravis G, Flechon A, Chevreau C, Mahammedi H, Laguerre B, Guillot A, Joly F, Soulie M, Allory Y, Harter V, Culine S; VESPER Trial Investigators. Dose-Dense Methotrexate, Vinblastine, Doxorubicin, and Cisplatin or Gemcitabine and Cisplatin as Perioperative Chemotherapy for Patients With Nonmetastatic Muscle-Invasive Bladder Cancer: Results of the GETUG-AFU V05 VESPER Trial. J Clin Oncol. 2022 Jun 20;40(18):2013-2022. doi: 10.1200/JCO.21.02051. Epub 2022 Mar 7. PMID 35254888
- [Background] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Background] Willigenburg T, de Muinck Keizer DM, Peters M, Claes A, Lagendijk JJW, de Boer HCJ, van der Voort van Zyp JRN. Evaluation of daily online contour adaptation by radiation therapists for prostate cancer treatment on an MRI-guided linear accelerator. Clin Transl Radiat Oncol. 2021 Jan 14;27:50-56. doi: 10.1016/j.ctro.2021.01.002. eCollection 2021 Mar. PMID 33532630
- [Background] Caffo O, Fellin G, Graffer U, Mussari S, Tomio L, Galligioni E. Gemcitabine and radiotherapy plus cisplatin after transurethral resection as conservative treatment for infiltrating bladder cancer: Long-term cumulative results of 2 prospective single-institution studies. Cancer. 2011 Mar 15;117(6):1190-6. doi: 10.1002/cncr.25667. Epub 2010 Oct 19. PMID 20960501
- [Background] Coppin CM, Gospodarowicz MK, James K, Tannock IF, Zee B, Carson J, Pater J, Sullivan LD. Improved local control of invasive bladder cancer by concurrent cisplatin and preoperative or definitive radiation. The National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 1996 Nov;14(11):2901-7. doi: 10.1200/JCO.1996.14.11.2901. PMID 8918486
- [Background] Gronborg C, Vestergaard A, Hoyer M, Sohn M, Pedersen EM, Petersen JB, Agerbaek M, Muren LP. Intra-fractional bladder motion and margins in adaptive radiotherapy for urinary bladder cancer. Acta Oncol. 2015;54(9):1461-6. doi: 10.3109/0284186X.2015.1062138. Epub 2015 Aug 27. PMID 26313410
- [Background] Giacalone NJ, Shipley WU, Clayman RH, Niemierko A, Drumm M, Heney NM, Michaelson MD, Lee RJ, Saylor PJ, Wszolek MF, Feldman AS, Dahl DM, Zietman AL, Efstathiou JA. Long-term Outcomes After Bladder-preserving Tri-modality Therapy for Patients with Muscle-invasive Bladder Cancer: An Updated Analysis of the Massachusetts General Hospital Experience. Eur Urol. 2017 Jun;71(6):952-960. doi: 10.1016/j.eururo.2016.12.020. Epub 2017 Jan 9. PMID 28081860
- [Background] Mak RH, Hunt D, Shipley WU, Efstathiou JA, Tester WJ, Hagan MP, Kaufman DS, Heney NM, Zietman AL. Long-term outcomes in patients with muscle-invasive bladder cancer after selective bladder-preserving combined-modality therapy: a pooled analysis of Radiation Therapy Oncology Group protocols 8802, 8903, 9506, 9706, 9906, and 0233. J Clin Oncol. 2014 Dec 1;32(34):3801-9. doi: 10.1200/JCO.2014.57.5548. Epub 2014 Nov 3. PMID 25366678
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524
- [Background] Shi H, Zhang W, Bi X, Wang D, Xiao Z, Guan Y, Guan K, Tian J, Bai H, Hu L, Cao C, Jiang W, Hu Z, Zhang J, Chen Y, Zheng S, Feng X, Li C, Li Y, Ma J, Liu Y, Zhou A, Shou J. Neoadjuvant Chemotherapy-Guided Bladder-Sparing Treatment for Muscle-Invasive Bladder Cancer: Results of a Pilot Phase II Study. Cancer Res Treat. 2021 Oct;53(4):1156-1165. doi: 10.4143/crt.2020.1356. Epub 2021 Feb 10. PMID 33592141
- [Background] Cho SW, Lim SH, Kwon GY, Kim CK, Park W, Pyo H, Chung JH, Song W, Sung HH, Jeong BC, Park SH. Neoadjuvant Cisplatin-Based Chemotherapy Followed by Selective Bladder Preservation Chemoradiotherapy in Muscle-Invasive Urothelial Carcinoma of the Bladder: Post Hoc Analysis of Two Prospective Studies. Cancer Res Treat. 2024 Jul;56(3):893-897. doi: 10.4143/crt.2024.015. Epub 2024 Feb 15. PMID 38374699
- [Background] Tester W, Caplan R, Heaney J, Venner P, Whittington R, Byhardt R, True L, Shipley W. Neoadjuvant combined modality program with selective organ preservation for invasive bladder cancer: results of Radiation Therapy Oncology Group phase II trial 8802. J Clin Oncol. 1996 Jan;14(1):119-26. doi: 10.1200/JCO.1996.14.1.119. PMID 8558186
- [Background] Astrom LM, Behrens CP, Calmels L, Sjostrom D, Geertsen P, Mouritsen LS, Serup-Hansen E, Lindberg H, Sibolt P. Online adaptive radiotherapy of urinary bladder cancer with full re-optimization to the anatomy of the day: Initial experience and dosimetric benefits. Radiother Oncol. 2022 Jun;171:37-42. doi: 10.1016/j.radonc.2022.03.014. Epub 2022 Mar 28. PMID 35358605
- [Background] Sangar VK, McBain CA, Lyons J, Ramani VA, Logue JP, Wylie JP, Clarke NW, Cowan RA. Phase I study of conformal radiotherapy with concurrent gemcitabine in locally advanced bladder cancer. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):420-5. doi: 10.1016/j.ijrobp.2004.05.074. PMID 15667962
- [Background] Caffo O, Fellin G, Graffer U, Valduga F, Bolner A, Luciani L, Tomio L, Galligioni E. Phase I study of gemcitabine and radiotherapy plus cisplatin after transurethral resection as conservative treatment for infiltrating bladder cancer. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1310-6. doi: 10.1016/s0360-3016(03)00763-6. PMID 14630267
- [Background] Borut K, Lijana ZK. Phase I study of radiochemotherapy with gemcitabine in invasive bladder cancer. Radiother Oncol. 2012 Mar;102(3):412-5. doi: 10.1016/j.radonc.2011.07.026. Epub 2011 Sep 2. PMID 21890225
- [Background] Choudhury A, Swindell R, Logue JP, Elliott PA, Livsey JE, Wise M, Symonds P, Wylie JP, Ramani V, Sangar V, Lyons J, Bottomley I, McCaul D, Clarke NW, Kiltie AE, Cowan RA. Phase II study of conformal hypofractionated radiotherapy with concurrent gemcitabine in muscle-invasive bladder cancer. J Clin Oncol. 2011 Feb 20;29(6):733-8. doi: 10.1200/JCO.2010.31.5721. Epub 2011 Jan 4. PMID 21205754
- [Background] Shipley WU, Winter KA, Kaufman DS, Lee WR, Heney NM, Tester WR, Donnelly BJ, Venner PM, Perez CA, Murray KJ, Doggett RS, True LD. Phase III trial of neoadjuvant chemotherapy in patients with invasive bladder cancer treated with selective bladder preservation by combined radiation therapy and chemotherapy: initial results of Radiation Therapy Oncology Group 89-03. J Clin Oncol. 1998 Nov;16(11):3576-83. doi: 10.1200/JCO.1998.16.11.3576. PMID 9817278
- [Background] McNair HA, Joyce E, O'Gara G, Jackson M, Peet B, Huddart RA, Wiseman T. Radiographer-led online image guided adaptive radiotherapy: A qualitative investigation of the therapeutic radiographer role. Radiography (Lond). 2021 Nov;27(4):1085-1093. doi: 10.1016/j.radi.2021.04.012. Epub 2021 May 15. PMID 34006442
- [Background] James ND, Hussain SA, Hall E, Jenkins P, Tremlett J, Rawlings C, Crundwell M, Sizer B, Sreenivasan T, Hendron C, Lewis R, Waters R, Huddart RA; BC2001 Investigators. Radiotherapy with or without chemotherapy in muscle-invasive bladder cancer. N Engl J Med. 2012 Apr 19;366(16):1477-88. doi: 10.1056/NEJMoa1106106. PMID 22512481
- [Background] Huddart RA, Hall E, Hussain SA, Jenkins P, Rawlings C, Tremlett J, Crundwell M, Adab FA, Sheehan D, Syndikus I, Hendron C, Lewis R, Waters R, James ND. Randomized noninferiority trial of reduced high-dose volume versus standard volume radiation therapy for muscle-invasive bladder cancer: results of the BC2001 trial (CRUK/01/004). Int J Radiat Oncol Biol Phys. 2013 Oct 1;87(2):261-9. doi: 10.1016/j.ijrobp.2013.06.2044. PMID 23958147
- [Background] Khalifa J, Supiot S, Pignot G, Hennequin C, Blanchard P, Pasquier D, Magne N, de Crevoisier R, Graff-Cailleaud P, Riou O, Cabaille M, Azria D, Latorzeff I, Crehange G, Chapet O, Roupret M, Belhomme S, Mejean A, Culine S, Sargos P. Recommendations for planning and delivery of radical radiotherapy for localized urothelial carcinoma of the bladder. Radiother Oncol. 2021 Aug;161:95-114. doi: 10.1016/j.radonc.2021.06.011. Epub 2021 Jun 10. PMID 34118357
- [Background] Amestoy F, Roubaud G, Antoine M, Fonteyne V, Baumann BC, Christodouleas J, Roupret M, Azria D, Zilli T, Hennequin C, Xylinas E, Sargos P; Young Academic Urologists Urothelial Carcinoma Group of the European Association of Urology. Review of hypo-fractionated radiotherapy for localized muscle invasive bladder cancer. Crit Rev Oncol Hematol. 2019 Oct;142:76-85. doi: 10.1016/j.critrevonc.2019.06.010. Epub 2019 Jul 16. PMID 31377435
- [Background] Fabiano E, Riou O, Pointreau Y, Perichon N, Durdux C. Role of radiotherapy in the management of bladder cancer: Recommendations of the French society for radiation oncology. Cancer Radiother. 2022 Feb-Apr;26(1-2):315-322. doi: 10.1016/j.canrad.2021.11.006. Epub 2021 Dec 23. PMID 34955411
- [Background] Reignier PL, Gauthier H, Hennequin C, Aussedat Q, Xylinas E, Desgrandchamps F, Culine S, Masson-Lecomte A, Dumont C. Survival after sequential neoadjuvant chemotherapy followed by trimodal treatment or radical cystectomy for muscle-invasive bladder cancer. World J Urol. 2023 Nov;41(11):3249-3255. doi: 10.1007/s00345-023-04506-9. Epub 2023 Jul 6. PMID 37410102
- [Background] Thompson C, Joseph N, Sanderson B, Logue J, Wylie J, Elliott T, Lyons J, Anandadas C, Choudhury A. Tolerability of Concurrent Chemoradiation Therapy With Gemcitabine (GemX), With and Without Prior Neoadjuvant Chemotherapy, in Muscle Invasive Bladder Cancer. Int J Radiat Oncol Biol Phys. 2017 Mar 15;97(4):732-739. doi: 10.1016/j.ijrobp.2016.11.040. Epub 2016 Nov 27. PMID 28244408
- See also: incidence et de la mortalité par cancer en France métropolitaine — https://www.santepubliquefrance.fr/maladies-et-traumatismes/cancers/cancer-du-sein/documents/rapport-synthese/estimations-nationales-de-l-incidence-et-de-la-mortalite-par-cancer-en-france-metropolitaine-entre-1990-et-2018-volume-1-tumeurs-solides-etud